CLINICAL TRIAL: NCT00241943
Title: Cooperative Agreement to Develop, Implement, and Evaluate Viral Hepatitis and Training
Brief Title: A Video-Based HCV Curriculum for Active Injection Drug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organization to Achieve Solutions in Substance Abuse (OASIS) (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Diana Sylvestre, MD, OASIS
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: U50/CCU923257-2; U50/CCU923257
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Hepatitis C; Opiate Dependence
Keywords: Hepatitis C; Heroin; Populations at risk; testing; vaccination
MeSH Terms: conditions — Hepatitis C; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Hepatitis C educational video

SUMMARY:
The investigators hypothesize that a well-designed hepatitis C (HCV) video education curriculum for active drug injectors will lead to measurable improvements in HCV testing rates, HAV and HBV vaccination rates, as well as knowledge and attitudes about this condition. The investigators will use a short 10 minute video designed for active drug users to and assess its impact vs. a usual-care counseling intervention. The investigators will measure and compare its impact at baseline, 4 weeks after video viewing, and 12 weeks after intervention.

DETAILED DESCRIPTION:
Active drug injectors are at high risk for contracting and transmitting HCV. Very few culturally-specific tools have been developed to improve outcomes in this population. We hypothesize that measurable improvements in HCV testing rates, hepatitis A and B vaccination rates, and knowledge, attitudes, and motivations toward behavior change may be elicited by such a curriculum.

In this study, we will investigate the impact of a short HCV education video on active drug injectors at a syringe exchange program. Subjects will be enrolled in one of two cohorts: a usual-care cohort, which will receive the program's standard HCV counseling; vs an intervention cohort, which will view the education video. Subjects will undergo written testing for knowledge, attitudes about transmission behaviors, and motivations toward behavior change before the intervention, immediately after the intervention, 4 weeks after the intervention, and 12 weeks after the intervention. Additionally, we will measure and compare the rates of HCV testing and HAV/HBV vaccinations before and at the end of the 12 week time point in both cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Attendance at syringe exchange program

Exclusion Criteria:

* Unable to provide informed consent
* Not interested in study
* Not able to speak or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
HCV testing rates, intervention vs. usual care
HAV vaccination rates, intervention vs. usual care
HBV vaccination rates, intervention vs. usual care

SECONDARY OUTCOMES:
Improvement in knowledge, intervention vs. usual care
Improvement in attitudes toward behavior change, intervention vs. usual care
Improvement in motivations toward behavior change, intervention vs. usual care

CONTACTS AND LOCATIONS:
Overall Officials: Diana L. Sylvestre, MD, Principal Investigator — Organization to Achieve Solutions in Substance Abuse (OASIS)
Locations (1):
- HEPPAC, Oakland, California, United States